CLINICAL TRIAL: NCT00938054
Title: Characterization of Autism Spectrum Disorder in School Aged Children
Brief Title: Identification of Characteristics Associated With Symptom Remission in Autism
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090171; 09-M-0171
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2012-10-09

CONDITIONS: Autism Spectrum Disorders; Autism
Keywords: Outcome; Autism; Pervasive Developmental Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Autism is defined as a lifelong pervasive developmental disability, as such, symptom recovery is considered rare. Reports by Lovaas and McEachin, Smith & Lovaas and more recently by Cohen, Amerine-Dickens, & Smith, Smith Groen et al. and Sutera Pandey et al suggest that intensive behavioral intervention programs during preschool years may result in improvement to the point where some children no longer meet criteria for autism by the time they reach school age. Similarly, there are a large number of anecdotal reports of children with autism who, following intensive biomedical intervention (e.g., gluten/casein free diets, vitamin supplements, chelation), are indistinguishable from their typically developing peers. The goal of the current research is to characterize the behavioral and biological profiles of children with autism who show significant symptom reduction such that they no longer meet criteria for autism (Remitted Autism [REM-AUT]) and to contrast them with a group of children who continue to meet criteria for autism (AUT) and to typically developing (TD) group of children. Examining whether neurobiological and neurobehavioral symptoms commonly reported in autism are as frequent and severe in children who have responded to treatment is an important first step in determining what factors may contribute to symptom remission in autism. In addition, understanding how children with remitted autism compare to typically developing children will help us better understand whether symptom improvement is through remediation (normalization of function) or compensation (achieving the same behavioral/adaptive outcome but through an alternative process).

DETAILED DESCRIPTION:
Autism is defined as a lifelong pervasive developmental disability, as such, symptom recovery is considered rare. Reports by Lovaas and McEachin, Smith & Lovaas and more recently by Cohen, Amerine-Dickens, & Smith, Smith Groen et al. and Sutera Pandey et al suggest that intensive behavioral intervention programs during preschool years may result in improvement to the point where some children no longer meet criteria for autism by the time they reach school age. Similarly, there are a large number of anecdotal reports of children with autism who, following intensive biomedical intervention (e.g., gluten/casein free diets, vitamin supplements, chelation), are indistinguishable from their typically developing peers. The goal of the current research is to characterize the behavioral and biological profiles of children with autism who show significant symptom reduction such that they no longer meet criteria for autism (Remitted Autism [REM-AUT]) and to contrast them with a group of children who continue to meet criteria for autism (AUT) and to typically developing (TD) group of children. Examining whether neurobiological and neurobehavioral symptoms commonly reported in autism are as frequent and severe in children who have responded to treatment is an important first step in determining what factors may contribute to symptom remission in autism. In addition, understanding how children with remitted autism compare to typically developing children will help us better understand whether symptom improvement is through remediation (normalization of function) or compensation (achieving the same behavioral/adaptive outcome but through an alternative process).

ELIGIBILITY:
* INCLUSION CRITERIA:

STUDY SUBJECTS:

Remitted Autism (REM-AUT) Group:

1. Diagnosis of autism prior to symptom improvement

   1. valid administration of ADI and/or ADOS with accompanying interpretive report yielding an autism diagnosis

      OR
   2. clinical/developmental evaluation including a detailed review of the child s history and direct observation of current behavioral functioning resulting in a documented diagnosis of autism by a child developmental specialist experienced with autism spectrum disorders such as a developmental pediatrician, developmental psychologist, child clinical psychologist, or a child psychiatrist
   3. measure of cognitive ability from within 1 year of initial autism diagnosis
   4. objective measure indicative of prominent autism symptoms using a recognized and standardized assessment of autism symptoms such as the Social Responsiveness Scale (SRS), Childhood Autism Rating Scale (CARS), or the Modified Checklist for Autism in Toddlers (MCHAT) or video tapes of assessments
   5. initial diagnosis of autism prior to age 6

      AND
   6. Medical, educational, treatment record review by PDN branch clinicians to confirm diagnostic impressions including a detailed description of child s behaviors that support an autism diagnosis
   7. The final decision for meeting diagnostic and treatment history inclusion criteria is based on PDN branch staff review of the case
   8. Treatment history: all participants must have received adequate treatment intervention for their autism symptoms. Participant medical and treatment records will be carefully reviewed to ascertain their treatment history
2. Current functioning:

   a. Parent report and report of at least one professional that child is no longer autistic
3. At screening visit (after meeting initial eligibility), will not meet criteria for autism

   1. Must not meet criteria for autism per overall clinical impression based on information collected from administration of the ADOS, current ADI-R symptoms, and other clinical observations made the assessment.
   2. Teacher/informant report of autism symptoms (such as results from the SRS) not indicative of autism diagnosis
   3. Minimum improvement of symptoms required from group assignment: approximately 2 point CGI severity of illness change (or equivalent) based on PDN impression of change in illness severity from initial diagnosis (estimated based on review of past medical records) and current functioning

      OR
   4. Current assessment of functional impairment due to autism symptoms using a standardized assessment measure such as the Developmental Disability-Children s Global Assessment Scale will reflect adequate functioning in all areas and/or a clinically significant improvement in functioning, consistent with common psychiatric treatment definitions for treatment response
4. Able to participate in study procedures.

AUTISM Group:

1. Diagnosis of autism following the same criteria as described above
2. Treatment history: all study participants must have received adequate treatment intervention. Treatment history will be matched to treatment provided to children in the REM-AUT group.
3. Screening visit (after meeting initial eligibility): will meet criteria for autistic disorder using the same diagnostic process described for the REM-AUT group above
4. Matched to REM-AUT group on IQ, age of diagnosis, and treatment history. IQ matching between the AUT and REM-AUT groups will be based on pretreatment estimates of cognitive level obtained from the medical record review.
5. Able to participate in study procedures.

TD Group:

1. IQ matched to a sub-sample of children in the REM-AUT group with normal range intellectual functioning. IQ matching between the TD and REM-AUT groups will be based on current intellectual functioning at the time of study participation.
2. Able to participate in study procedures.

EXCLUSION CRITERIA:

All groups: May not be pregnant or have a known genetic disorder, mitochondrial disease, history of birth trauma, or current uncontrolled seizures

TD Group:

1. Current diagnosis or significant history of pervasive developmental disorder, language delay or disorder (except articulation), attention or learning issues, or major psychiatric condition.
2. Prematurity at birth less than 36 weeks gestation); or birth weight significantly below normal for gestational age (SGA- small for gestational age).

PARENTS OF ALL STUDY PARTICIPANTS:

As noted parents of all study groups will provide DNA, plasma, and serum samples.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-06-25; Study Completion 2012-10-09

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abrahams BS, Geschwind DH. Advances in autism genetics: on the threshold of a new neurobiology. Nat Rev Genet. 2008 May;9(5):341-55. doi: 10.1038/nrg2346. PMID 18414403
- [Background] Bibby P, Eikeseth S, Martin NT, Mudford OC, Reeves D. Progress and outcomes for children with autism receiving parent-managed intensive interventions. Res Dev Disabil. 2002 Jan-Feb;23(1):81-104. doi: 10.1016/s0891-4222(02)00095-1. PMID 12071397
- [Background] Boyd RD, Corley MJ. Outcome survey of early intensive behavioral intervention for young children with autism in a community setting. Autism. 2001 Dec;5(4):430-41. doi: 10.1177/1362361301005004007. PMID 11777258